CLINICAL TRIAL: NCT03311841
Title: A Study to Assess the Pharmacokinetics of Midazolam, Dabigatran, Pitavastatin, Atorvastatin, and Rosuvastatin Administered as Microdoses in Subjects With Varying Degrees of Renal Insufficiency in the Presence and Absence of Rifampin
Brief Title: Pharmacokinetics of Midazolam, Dabigatran, Pitavastatin, Atorvastatin, and Rosuvastatin in Participants With Renal Insufficiency in the Presence and Absence of Rifampin (MK-0000-386)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000-386; MK-0000-386 (Other: Merck); CA21005 (Other: Celerion)
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Midazolam; Dabigatran; pitavastatin; Atorvastatin; Rosuvastatin Calcium; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- End Stage Renal Disease (Experimental): Participants requiring hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). A washout period of at least 14 days will separate dosings.
  Interventions: Drug: Midazolam oral solution; Drug: Dabigatran and pitavastatin oral solution; Drug: Atorvastatin and rosuvastatin oral solution
- Severe Impairment (Experimental): Participants with <30 mL/min/1.73m^2 estimated glomerular filtration rate (eGFR) not on hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
  Interventions: Drug: Midazolam oral solution; Drug: Dabigatran and pitavastatin oral solution; Drug: Atorvastatin and rosuvastatin oral solution; Drug: Rifampin
- Moderate Impairment (Experimental): Participants with 30 to <60 mL/min/1.73m^2 eGFR not on hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
  Interventions: Drug: Midazolam oral solution; Drug: Dabigatran and pitavastatin oral solution; Drug: Atorvastatin and rosuvastatin oral solution; Drug: Rifampin
- Mild Impairment (Experimental): Participants with 60 to <90 mL/min/1.73m^2 eGFR not on hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
  Interventions: Drug: Midazolam oral solution; Drug: Dabigatran and pitavastatin oral solution; Drug: Atorvastatin and rosuvastatin oral solution; Drug: Rifampin
- Healthy Control (Active Comparator): Participants with ≥90 mL/min creatinine clearance. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
  Interventions: Drug: Midazolam oral solution; Drug: Dabigatran and pitavastatin oral solution; Drug: Atorvastatin and rosuvastatin oral solution; Drug: Rifampin

INTERVENTIONS:
Drug: Midazolam oral solution — Midazolam hydrochloride 10 μg (1 mL of 10 μg/mL oral solution), administered orally as part of a microdose cocktail
Drug: Dabigatran and pitavastatin oral solution — 375/10 μg dabigatran etexilate and pitavastatin (1 mL of 375/10 μg/mL oral solution), administered orally as part of a microdose cocktail
Drug: Atorvastatin and rosuvastatin oral solution — 100/50 μg atorvastatin and rosuvastatin (2 mL of 50/25 μg/mL oral solution), administered orally as part of a microdose cocktail
Drug: Rifampin — Rifampin 600 mg single dose (two 300 mg capsules) administered orally
  Arms: Healthy Control; Mild Impairment; Moderate Impairment; Severe Impairment

SUMMARY:
The purpose of this open-label, 2-period, fixed-sequence study is to characterize the plasma pharmacokinetic profiles of midazolam, dabigatran, pitavastatin, atorvastatin, and rosuvastatin following a single oral dose administration of a microdose cocktail in healthy participants, in participants with mild, moderate, severe (not on dialysis) renal impairment, and in participants with end-stage renal disease (ESRD; on dialysis).

ELIGIBILITY:
Inclusion Criteria:

All participants (with mild, moderate or severe renal impairment, end stage renal disease, or healthy):

* a female must be non-pregnant, non-breast feeding and if she is of reproductive potential: must agree to use (and/or have their partner use) two acceptable methods of birth control beginning at screening, throughout the study and until 2 weeks after the last dosing of study drug
* a female of non-childbearing potential: must have undergone a sterilization procedure at least 6 months prior to the first dose or be postmenopausal with amenorrhea for at least 1 year prior to the first dose
* a non-vasectomized male participant must agree to use a condom with spermicide or abstain from sexual intercourse from the first dose until 90 days after the last dose of study drug
* a male participant must agree not to donate sperm from dosing until 90 days after the last dose of study drug
* has a body mass index (BMI) ≤ 40.0 kg/m^2
* is a non-smoker or moderate smoker (≤ 20 cigarettes/day or the equivalent)

Participants with mild, moderate or severe renal impairment or end stage renal disease:

* has a clinical diagnosis of renal impairment and meets the protocol-specified renal impairment function qualifications at the prestudy visit (screening)

Healthy participants:

* has baseline creatinine clearance ≥ 90 mL/min based on Cockcroft-Gault equation
* is judged to be in good health based on medical history, physical examination, vital signs, pulse oximetry, and laboratory safety tests

Exclusion Criteria:

All participants (with mild, moderate or severe renal impairment, end stage renal disease, or healthy):

* is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* history or presence of clinically significant medical or psychiatric condition or disease
* history of stroke, chronic seizures, or major neurological disorders
* history of malignant neoplastic disease
* history or presence of alcoholism or drug abuse within the past 6 months
* female participant who is pregnant or lactating

Participants with mild, moderate or severe renal impairment:

* has had a renal transplant or has had nephrectomy
* has uncontrolled type 2 diabetes mellitus (T2DM), a history of Type 1 diabetes, or ketoacidosis
* history of significant endocrine, gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary diseases

Participants with end stage renal disease (ESRD):

* had a failed renal allograft within the last 2 years prior to the first dose, or a successful renal allograft
* has uncontrolled T2DM, a history of Type 1 diabetes, or ketoacidosis
* history of significant endocrine, gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary diseases

Healthy participants:

* history of hypoglycemia, glucose intolerance, T2DM, or ketoacidosis
* history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami ( Site 0001), Hialeah, Florida
  - Orlando Clinical Research Center ( Site 0002), Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- End-Stage Renal Disease: Participants requiring hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). A washout period of at least 14 days will separate dosings
Period: Period 1
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Started | 6 | 7 | 6 | 7 | 6
Completed | 6 | 7 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 14-day Wash-out
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Started | 6 | 7 | 6 | 7 | 6
Completed | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Started | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control | Total
Number analyzed (Participants) | 6 | 7 | 6 | 7 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (8.04) | 64.9 (7.10) | 67.0 (11.19) | 65.4 (8.90) | 57.8 (7.88) | 62.5 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 3 | 3 | 11
  Male | 6 | 6 | 2 | 4 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 4 | 5 | 6 | 20
  Not Hispanic or Latino | 6 | 2 | 2 | 2 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 00 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 0 | 0 | 3 | 0 | 9
  White | 0 | 7 | 6 | 3 | 6 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) Post-dose Period 1
Description: AUC0-inf is the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease (ESRD) requiring hemodialysis.
Time Frame: 0 hour (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of AUC0-inf for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg*hr/mL
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
pg*hr/mL
  Midazolam | 110 [74.6 to 162] | 260 [181 to 372] | 364 [247 to 537] | 176 [119 to 259] | 273 [185 to 403]
  Dabigatran: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Dabigatran | 5370 [3410 to 8460] | 7900 [5010 to 12400] | 4550 [2890 to 7180] | 1610 [1020 to 2530] | 1580 [1010 to 2500]
  Pitavastatin | 676 [456 to 1000] | 648 [450 to 933] | 1020 [686 to 1510] | 688 [464 to 1020] | 520 [350 to 771]
  Pitavastatin lactone (metabolite) | 1100 [774 to 1560] | 1680 [1220 to 2320] | 2240 [1580 to 3170] | 1610 [1140 to 2290] | 1540 [1090 to 2190]
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 329 [203 to 531] | 476 [305 to 743] | 511 [316 to 826] | 329 [183 to 593] | 292 [180 to 472]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 6 | 7 | 5 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) | 163 [112 to 237] | 226 [160 to 319] | 273 [181 to 411] | 286 [181 to 453] | 208 [143 to 302]
  Rosuvastatin: number analyzed (Participants) | 5 | 6 | 5 | 4 | 3
  Rosuvastatin | 208 [116 to 374] | 365 [213 to 624] | 575 [319 to 1030] | 262 [136 to 505] | 292 [137 to 624]
Statistical Analysis 1: Comparison: Mild Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.64, 95% CI 2-sided [0.37 to 1.11] — Geometric least squares mean ratio and 95% confidence interval could not be determined for comparisons where one or both of the geometric least squares means was not calculable because some individual values were treated as 0
Statistical Analysis 2: Comparison: Moderate Impairment vs Healthy Control; Comparison of midazolam; Test type: Other — Geometric least squares mean ratio and 95% confidence interval could not be determined for comparisons where one or both of the geometric least squares means was not calculable because some individual values were treated as 0; Geometric least squares mean ratio = 1.33, 95% CI 2-sided [0.77 to 2.31]
Statistical Analysis 3: Comparison: Severe Impairment vs Healthy Control; Comparison of midazolam; Test type: Other — [test comment as in outcome 1, analysis 2]; Geometric least squares mean ratio = 0.95, 95% CI 2-sided [0.56 to 1.62]
Statistical Analysis 4: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.40, 95% CI 2-sided [0.23 to 0.70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Mild Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 1.01, 95% CI 2-sided [0.53 to 1.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Moderate Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 2.87, 95% CI 2-sided [1.51 to 5.47] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Severe Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 4.98, 95% CI 2-sided [2.62 to 9.48] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 3.39, 95% CI 2-sided [1.78 to 6.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Mild Impairment vs Healthy Control; Test type: Other — Comparison of pitavastatin; Geometric least squares mean ratio = 1.32, 95% CI 2-sided [0.76 to 2.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.96, 95% CI 2-sided [1.12 to 3.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.25, 95% CI 2-sided [0.73 to 2.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.30, 95% CI 2-sided [0.74 to 2.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.05, 95% CI 2-sided [0.64 to 1.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.45, 95% CI 2-sided [0.88 to 2.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Severe Impairment vs Healthy Control; Test type: Other — Comparison of pitavastatin lactone; Geometric least squares mean ratio = 1.09, 95% CI 2-sided [0.68 to 1.76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: End-Stage Renal Disease vs Healthy Control; Test type: Other — Comparison of pitavastatin lactone; Geometric least squares mean ratio = 0.71, 95% CI 2-sided [0.43 to 1.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Mild Impairment vs Healthy Control; Test type: Other — Comparison of atorvastatin; Geometric least squares mean ratio = 1.13, 95% CI 2-sided [0.53 to 2.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Moderate Impairment vs Healthy Control; Test type: Other — Comparison of atorvastatin; Geometric least squares mean ratio = 1.75, 95% CI 2-sided [0.89 to 3.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Severe Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.63, 95% CI 2-sided [0.85 to 3.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: End-Stage Renal Disease vs Healthy Control; Test type: Other — Comparison of atorvastatin; Geometric least squares mean ratio = 1.13, 95% CI 2-sided [0.57 to 2.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Mild Impairment vs Healthy Control; Test type: Other — Comparison of ortho-hydroxyatorvastatin; Geometric least squares mean ratio = 1.38, 95% CI 2-sided [0.76 to 2.49] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Moderate Impairment vs Healthy Control; Test type: Other — Comparison of ortho-hydroxyatorvastatin; Geometric least squares mean ratio = 1.31, 95% CI 2-sided [0.75 to 2.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Severe Impairment vs Healthy Control; Test type: Other — Comparison of ortho-hydroxyatorvastatin; Geometric least squares mean ratio = 1.09, 95% CI 2-sided [0.65 to 1.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: End-Stage Renal Disease vs Healthy Control; Test type: Other — Comparison of ortho-hydroxyatorvastatin; Geometric least squares mean ratio = 0.79, 95% CI 2-sided [0.46 to 1.33] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Mild Impairment vs Healthy Control; Test type: Other — Comparison of rosuvastatin; Geometric least squares mean ratio = 0.90, 95% CI 2-sided [0.33 to 2.45] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: Moderate Impairment vs Healthy Control; Test type: Other — Comparison of rosuvastatin; Geometric least squares mean ratio = 1.97, 95% CI 2-sided [0.75 to 5.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: Severe Impairment vs Healthy Control; Test type: Other — Comparison of rosuvastatin; Geometric least squares mean ratio = 1.25, 95% CI 2-sided [0.49 to 3.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: End-Stage Renal Disease vs Healthy Control; Test type: Other — Comparison of rosuvastatin; Geometric least squares mean ratio = 0.71, 95% CI 2-sided [0.27 to 1.86] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Effect of Rifampin on AUC0-inf Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the AUC0-inf of midazolam, dabigatran, pitavastatin, pitavastatin lactone, atorvastatin, ortho-hydroxyatorvastatin, and rosuvatatin. AUC0-inf is the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include data from the end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: Microdose cocktail: 0 hour (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose; rifampin: 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 24 hours post-dose
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of AUC0-inf for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg*hr/mL
Groups:
- End Stage Renal Disease (Period 2): Participants requiring hemodialysis. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution).
- Severe Impairment (Period 2): Participants with <30 mL/min/1.73m^2 estimated glomerular filtration rate (eGFR) not on hemodialysis. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin.
- Moderate Impairment (Period 2): Participants with 30 to <60 mL/min/1.73m^2 eGFR not on hemodialysis. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin.
- Mild Impairment (Period 2): Participants with 60 to <90 mL/min/1.73m^2 eGFR not on hemodialysis. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin.
- Healthy Control (Period 2): Participants with ≥90 mL/min creatinine clearance. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin.
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
pg*hr/mL
  Midazolam |  | 244 [175 to 340] | 359 [252 to 512] | 189 [132 to 269] | 239 [168 to 341]
  Dabigatran |  | 10700 [7390 to 15600] | 7240 [4990 to 10500] | 3040 [2090 to 4400] | 3290 [2270 to 4770]
  Pitavastatin |  | 2850 [1840 to 4440] | 3500 [2200 to 5570] | 2530 [1590 to 4030] | 1910 [1200 to 3030]
  Pitavastatin lactone (metabolite) |  | 1560 [1160 to 2100] | 2500 [1830 to 3430] | 1930 [1410 to 2640] | 1340 [981 to 1840]
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 2240 [1520 to 3320] | 2430 [1620 to 3650] | 1710 [1040 to 2810] | 1770 [1180 to 2660]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) |  | 1620 [1080 to 2430] | 1870 [1230 to 2840] | 1760 [1060 to 2940] | 1650 [1080 to 2500]
  Rosuvastatin: number analyzed (Participants) | 0 | 5 | 4 | 5 | 5
  Rosuvastatin |  | 1240 [839 to 1830] | 1800 [1150 to 2820] | 1060 [695 to 1620] | 830 [553 to 1250]

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC0-24) Post-dose Period 1
Description: AUC0-24 is the area under the plasma concentration-time curve from time 0 to 24 hours post-dose. This is a measure of the average amount of study drug in the blood plasma over a period of 24 hours after the dose. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease requiring hemodialysis.
Time Frame: 0 hour (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of AUC0-24 for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Mean (95% Confidence Interval); unit: pg*hr/mL
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
pg*hr/mL
  Midazolam | 106 [74.2 to 152] | 235 [169 to 328] | 317 [222 to 454] | 168 [117 to 240] | 252 [176 to 360]
  Dabigatran | 2100 [1380 to 3200] | 4470 [3030 to 6590] | 3440 [2260 to 5240] | 1380 [907 to 2100] | 1440 [949 to 2200]
  Pitavastatin | 593 [411 to 857] | 525 [374 to 738] | 764 [529 to 1100] | 543 [376 to 783] | 415 [288 to 600]
  Pitavastatin lactone (metabolite) | 858 [639 to 1150] | 1100 [835 to 1440] | 1280 [950 to 1710] | 1040 [772 to 1390] | 1010 [750 to 1350]
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 287 [184 to 446] | 300 [199 to 452] | 329 [211 to 512] | 219 [128 to 377] | 198 [127 to 308]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) | 115 [78.3 to 168] | 112 [78.5 to 159] | 143 [98.0 to 210] | 139 [86.9 to 221] | 108 [73.8 to 158]
  Rosuvastatin: number analyzed (Participants) | 6 | 7 | 6 | 5 | 6
  Rosuvastatin | 162 [97.2 to 271] | 223 [139 to 358] | 343 [206 to 573] | 191 [109 to 334] | 153 [91.6 to 255]
Statistical Analysis 1: Comparison: Mild Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.67, 95% CI 2-sided [0.40 to 1.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 1.26, 95% CI 2-sided [0.76 to 2.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.93, 95% CI 2-sided [0.57 to 1.52] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.42, 95% CI 2-sided [0.25 to 0.70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Mild Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 0.96, 95% CI 2-sided [0.53 to 1.73] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Moderate Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 2.38, 95% CI 2-sided [1.32 to 4.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Severe Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 3.09, 95% CI 2-sided [1.75 to 5.48] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 1.46, 95% CI 2-sided [0.80 to 2.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.31, 95% CI 2-sided [0.78 to 2.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.84, 95% CI 2-sided [1.09 to 3.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.26, 95% CI 2-sided [0.77 to 2.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.43, 95% CI 2-sided [0.85 to 2.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.03, 95% CI 2-sided [0.68 to 1.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.27, 95% CI 2-sided [0.83 to 1.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.09, 95% CI 2-sided [0.73 to 1.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 0.85, 95% CI 2-sided [0.56 to 1.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Mild Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.11, 95% CI 2-sided [0.55 to 2.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Moderate Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.66, 95% CI 2-sided [0.89 to 3.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Severe Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.52, 95% CI 2-sided [0.83 to 2.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.45, 95% CI 2-sided [0.78 to 2.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Mild Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.28, 95% CI 2-sided [0.70 to 2.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Moderate Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.33, 95% CI 2-sided [0.78 to 2.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Severe Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.03, 95% CI 2-sided [0.62 to 1.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.06, 95% CI 2-sided [0.62 to 1.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Mild Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.25, 95% CI 2-sided [0.58 to 2.67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: Moderate Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 2.25, 95% CI 2-sided [1.09 to 4.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: Severe Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.46, 95% CI 2-sided [0.72 to 2.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.06, 95% CI 2-sided [0.51 to 2.19] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Last (AUC0-last) Post-dose Period 1
Description: AUC0-last is the area under the plasma concentration-time curve from time zero to time of last measurable concentration. This is a measure of the amount of study drug in the blood plasma from pre-dose until the last measurable concentration of study drug could be determined. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease requiring hemodialysis.
Time Frame: 0 hour (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of AUC0-last for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Mean (95% Confidence Interval); unit: pg*hr/mL
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
pg*hr/mL
  Midazolam | 105 [70.8 to 156] | 248 [172 to 358] | 344 [232 to 511] | 167 [113 to 248] | 264 [178 to 392]
  Dabigatran | 3740 [2370 to 5910] | 7450 [4870 to 11400] | 4230 [2680 to 6690] | 1440 [910 to 2270] | 1410 [891 to 2230]
  Pitavastatin | 649 [435 to 968] | 602 [416 to 871] | 950 [637 to 1420] | 643 [431 to 959] | 483 [324 to 721]
  Pitavastatin lactone (metabolite) | 1060 [754 to 1480] | 1570 [1150 to 2140] | 2020 [1440 to 2830] | 1490 [1060 to 2080] | 1450 [1030 to 2030]
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 298 [182 to 488] | 419 [266 to 662] | 459 [280 to 751] | 295 [161 to 539] | 255 [155 to 417]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) | 126 [80.3 to 198] | 176 [116 to 267] | 256 [163 to 402] | 221 [127 to 385] | 152 [96.8 to 239]
  Rosuvastatin: number analyzed (Participants) | 6 | 7 | 6 | 5 | 6
  Rosuvastatin | 171 [98.0 to 298] | 269 [161 to 451] | 479 [274 to 835] | 231 [125 to 424] | 181 [104 to 315]
Statistical Analysis 1: Comparison: Mild Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.63, 95% CI 2-sided [0.36 to 1.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 1.30, 95% CI 2-sided [0.75 to 2.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.94, 95% CI 2-sided [0.55 to 1.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.40, 95% CI 2-sided [0.23 to 0.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Mild Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 1.02, 95% CI 2-sided [0.53 to 1.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Moderate Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 3.00, 95% CI 2-sided [1.57 to 5.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Severe Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 5.28, 95% CI 2-sided [2.83 to 9.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 2.65, 95% CI 2-sided [1.39 to 5.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.33, 95% CI 2-sided [0.76 to 2.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.97, 95% CI 2-sided [1.12 to 3.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.25, 95% CI 2-sided [0.72 to 2.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.34, 95% CI 2-sided [0.76 to 2.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.03, 95% CI 2-sided [0.64 to 1.65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.39, 95% CI 2-sided [0.87 to 2.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.08, 95% CI 2-sided [0.68 to 1.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 0.73, 95% CI 2-sided [0.45 to 1.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Mild Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.16, 95% CI 2-sided [0.53 to 2.52] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Moderate Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.80, 95% CI 2-sided [0.90 to 3.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Severe Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.65, 95% CI 2-sided [0.84 to 3.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.17, 95% CI 2-sided [0.58 to 2.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Mild Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.46, 95% CI 2-sided [0.71 to 2.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Moderate Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.68, 95% CI 2-sided [0.89 to 3.19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Severe Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.16, 95% CI 2-sided [0.63 to 2.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 0.83, 95% CI 2-sided [0.44 to 1.57] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Mild Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.27, 95% CI 2-sided [0.56 to 2.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: Moderate Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 2.65, 95% CI 2-sided [1.21 to 5.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: Severe Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.49, 95% CI 2-sided [0.70 to 3.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 0.95, 95% CI 2-sided [0.43 to 2.08] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Maximum Plasma Concentration (Cmax) Post-dose Period 1
Description: Cmax is the peak plasma concentration of study drug after administration. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease requiring hemodialysis.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of Cmax for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
pg/mL
  Midazolam | 39.9 [29.5 to 53.9] | 68.4 [51.8 to 90.4] | 77.2 [57.1 to 104] | 70.7 [52.3 to 95.5] | 73.2 [54.1 to 98.8]
  Dabigatran | 132 [83.1 to 208] | 319 [209 to 489] | 312 [197 to 494] | 153 [96.9 to 243] | 183 [115 to 290]
  Pitavastatin | 242 [173 to 339] | 218 [160 to 299] | 303 [216 to 425] | 244 [174 to 342] | 164 [117 to 230]
  Pitavastatin lactone (metabolite) | 78.5 [59.8 to 103] | 95.4 [74.2 to 123] | 106 [80.6 to 139] | 105 [79.9 to 137] | 88.1 [67.1 to 116]
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 63.7 [35.3 to 115] | 46.7 [27.1 to 80.5] | 55.0 [30.5 to 99.1] | 31.9 [15.5 to 65.7] | 21.6 [12.0 to 38.9]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) | 8.58 [5.77 to 12.8] | 7.22 [5.00 to 10.4] | 9.50 [6.39 to 14.1] | 8.50 [5.23 to 13.8] | 7.67 [5.16 to 11.4]
  Rosuvastatin: number analyzed (Participants) | 6 | 7 | 6 | 5 | 6
  Rosuvastatin | 22.5 [12.4 to 40.6] | 24.4 [14.1 to 42.1] | 40.4 [22.4 to 72.9] | 23.6 [12.4 to 45.1] | 21.5 [11.9 to 38.9]
Statistical Analysis 1: Comparison: Mild Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.97, 95% CI 2-sided [0.63 to 1.48] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Moderate Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 1.06, 95% CI 2-sided [0.69 to 1.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Severe Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.94, 95% CI 2-sided [0.62 to 1.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 0.55, 95% CI 2-sided [0.36 to 0.83] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Mild Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 0.84, 95% CI 2-sided [0.44 to 1.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Moderate Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 1.71, 95% CI 2-sided [0.89 to 3.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Severe Impairment vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 1.75, 95% CI 2-sided [0.93 to 3.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of dabigatran; Test type: Other; Geometric least squares mean ratio = 0.72, 95% CI 2-sided [0.38 to 1.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.49, 95% CI 2-sided [0.92 to 2.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.84, 95% CI 2-sided [1.14 to 2.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.33, 95% CI 2-sided [0.84 to 2.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.47, 95% CI 2-sided [0.91 to 2.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.19, 95% CI 2-sided [0.81 to 1.75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.20, 95% CI 2-sided [0.82 to 1.76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.08, 95% CI 2-sided [0.75 to 1.57] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 0.89, 95% CI 2-sided [0.61 to 1.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Mild Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 1.48, 95% CI 2-sided [0.58 to 3.75] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Moderate Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 2.54, 95% CI 2-sided [1.11 to 5.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Severe Impairment vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 2.16, 95% CI 2-sided [0.97 to 4.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of atorvastatin; Test type: Other; Geometric least squares mean ratio = 2.94, 95% CI 2-sided [1.28 to 6.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Mild Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.11, 95% CI 2-sided [0.59 to 2.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Moderate Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.24, 95% CI 2-sided [0.71 to 2.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Severe Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 0.94, 95% CI 2-sided [0.55 to 1.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.12, 95% CI 2-sided [0.64 to 1.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Mild Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.10, 95% CI 2-sided [0.46 to 2.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: Moderate Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.87, 95% CI 2-sided [0.81 to 4.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: Severe Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.13, 95% CI 2-sided [0.51 to 2.53] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.04, 95% CI 2-sided [0.45 to 2.41] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Plasma Concentration at 24 Hours (C24) Post-dose Period 1
Description: C24hr is a measure of the plasma study drug concentration 24 hours post-dose. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease requiring hemodialysis.
Time Frame: 24 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of C24 for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
pg/mL
  Midazolam | 0.283 [0.00 to 0.928] | 1.83 [0.00 to 8.47] | 2.64 [1.54 to 4.54] | 0.734 [0.00 to 1.06] | 1.57 [0.914 to 2.70]
  Dabigatran | 70.2 [45.3 to 109] | 107 [71.7 to 161] | 59.3 [38.3 to 91.8] | 18.7 [12.1 to 28.9] | 7.70 [0.00 to 26.6]
  Pitavastatin | 6.07 [0.00 to 7.99] | 4.04 [2.83 to 5.76] | 8.13 [5.53 to 11.9] | 5.32 [3.62 to 7.82] | 4.10 [2.79 to 6.03]
  Pitavastatin lactone (metabolite) | 12.9 [8.01 to 20.9] | 23.2 [14.9 to 36.2] | 32.8 [20.3 to 52.9] | 22.4 [13.9 to 36.2] | 21.7 [13.5 to 35.0]
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 4.28 [0.00 to 6.63] | 5.73 [3.80 to 8.64] | 6.03 [3.86 to 9.40] | 5.04 [2.73 to 5.89] | 3.85 [2.47 to 6.00]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) | 3.67 [0.00 to 4.64] | 3.25 [2.29 to 4.63] | 4.43 [3.03 to 6.49] | 5.02 [2.26 to 9.31] | 3.08 [2.10 to 4.51]
  Rosuvastatin: number analyzed (Participants) | 6 | 7 | 6 | 5 | 6
  Rosuvastatin | 2.64 [0.00 to 4.36] | 3.40 [2.24 to 5.16] | 6.01 [3.83 to 9.43] | 3.59 [2.19 to 5.88] | 1.94 [1.24 to 3.05]
Statistical Analysis 1: Comparison: Moderate Impairment vs Healthy Control; Comparison of midazolam; Test type: Other; Geometric least squares mean ratio = 1.68, 95% CI 2-sided [0.78 to 3.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.30, 95% CI 2-sided [0.75 to 2.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 1.98, 95% CI 2-sided [1.15 to 3.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin; Test type: Other; Geometric least squares mean ratio = 0.98, 95% CI 2-sided [0.58 to 1.66] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Mild Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.03, 95% CI 2-sided [0.52 to 2.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Moderate Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.51, 95% CI 2-sided [0.77 to 2.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Severe Impairment vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 1.07, 95% CI 2-sided [0.56 to 2.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: End-Stage Renal Disease vs Healthy Control; Comparison of pitavastatin lactone; Test type: Other; Geometric least squares mean ratio = 0.60, 95% CI 2-sided [0.30 to 1.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Moderate Impairment vs Healthy Control; Comparison of atovastatin; Test type: Other; Geometric least squares mean ratio = 1.57, 95% CI 2-sided [0.84 to 2.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Severe Impairment vs Healthy Control; Comparison of atovastatin; Test type: Other; Geometric least squares mean ratio = 1.49, 95% CI 2-sided [0.81 to 2.73] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Moderate Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.44, 95% CI 2-sided [0.84 to 2.47] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Severe Impairment vs Healthy Control; Comparison of ortho-hydroxyatorvastatin; Test type: Other; Geometric least squares mean ratio = 1.06, 95% CI 2-sided [0.63 to 1.78] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Mild Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.85, 95% CI 2-sided [0.95 to 3.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Moderate Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 3.10, 95% CI 2-sided [1.64 to 5.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Severe Impairment vs Healthy Control; Comparison of rosuvastatin; Test type: Other; Geometric least squares mean ratio = 1.75, 95% CI 2-sided [0.95 to 3.24] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) Post-dose Period 1
Description: Tmax is the amount of time to reach maximum (peak) plasma drug concentration following drug administration. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease requiring hemodialysis.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of Tmax for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
hours
  Midazolam | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 1.00 [0.50 to 1.00]
  Dabigatran | 2.00 [1.00 to 4.00] | 3.00 [2.00 to 4.00] | 2.50 [2.00 to 3.00] | 1.50 [1.50 to 3.00] | 1.50 [1.50 to 3.00]
  Pitavastatin | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.50] | 1.00 [0.50 to 1.00] | 0.52 [0.50 to 1.00] | 0.75 [0.50 to 1.00]
  Pitavastatin lactone (metabolite) | 2.50 [2.00 to 6.33] | 4.00 [2.00 to 4.00] | 2.50 [2.00 to 3.00] | 2.00 [1.50 to 2.00] | 2.00 [2.00 to 3.00]
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 0.25 [0.25 to 0.50] | 0.25 [0.25 to 6.00] | 0.25 [0.25 to 1.50] | 0.25 [0.25 to 0.53] | 0.50 [0.50 to 6.00]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) | 5.00 [4.00 to 6.00] | 6.00 [4.00 to 8.00] | 6.00 [4.00 to 8.00] | 6.00 [6.00 to 8.00] | 6.00 [3.00 to 6.00]
  Rosuvastatin: number analyzed (Participants) | 6 | 7 | 6 | 5 | 6
  Rosuvastatin | 3.00 [1.50 to 4.00] | 4.00 [3.00 to 4.00] | 4.00 [1.50 to 4.02] | 2.00 [2.00 to 4.00] | 3.50 [0.50 to 4.00]

8. Primary Outcome: Apparent Plasma Terminal Half-life (t1/2) Post-dose Period 1
Description: T1/2 is the elimination half-life of study drug. T1/2 is the time it takes for half of the study drug in the blood plasma to dissipate. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease requiring hemodialysis.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of t1/2 for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
hours
  Midazolam | 4.41 (59.6) | 7.79 (54.1) | 10.3 (33.0) | 6.76 (30.6) | 7.99 (25.0)
  Dabigatran: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Dabigatran | 41.4 (47.9) | 24.0 (22.0) | 11.9 (30.3) | 8.40 (10.7) | 6.75 (19.8)
  Pitavastatin | 11.8 (61.4) | 20.4 (63.6) | 22.4 (15.8) | 19.3 (23.5) | 17.8 (26.7)
  Pitavastatin lactone (metabolite) | 11.0 (55.3) | 18.1 (31.0) | 22.0 (13.2) | 20.5 (31.4) | 18.5 (15.9)
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 8.03 (28.5) | 17.5 (57.0) | 18.6 (41.8) | 16.7 (14.8) | 14.9 (10.3)
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 6 | 7 | 5 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) | 12.4 (25.8) | 21.9 (65.9) | 24.6 (18.3) | 22.8 (35.7) | 21.2 (29.5)
  Rosuvastatin: number analyzed (Participants) | 5 | 6 | 5 | 4 | 3
  Rosuvastatin | 14.0 (107.3) | 18.8 (78.3) | 24.9 (19.4) | 15.5 (100.2) | 16.2 (78.6)

9. Primary Outcome: Apparent Clearance After Extravascular Administration (CL/F) Post-dose Period 1
Description: CL/F is the rate at which study drug was removed from the body. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease requiring hemodialysis. CL/F was to be calculated for the parent plasma analytes only, midazolam, dabigatran, pitavastatin, atorvastatin, and rosuvastatin.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of CL/F for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
liters/hour
  Midazolam | 90.8 (46.5) | 38.5 (62.7) | 27.5 (46.3) | 56.9 (32.3) | 36.6 (50.6)
  Dabigatran: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Dabigatran | 52.5 (74.1) | 35.7 (32.3) | 61.8 (70.3) | 175 (47.3) | 178 (61.5)
  Pitavastatin | 14.8 (60.0) | 15.4 (58.6) | 9.84 (29.7) | 14.5 (41.1) | 19.2 (52.7)
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 304 (64.7) | 210 (82.9) | 196 (54.0) | 304 (28.7) | 343 (56.9)
  Rosuvastatin: number analyzed (Participants) | 5 | 6 | 5 | 4 | 3
  Rosuvastatin | 240 (121.0) | 137 (49.0) | 87.0 (32.3) | 191 (82.5) | 171 (47.8)

10. Primary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F) Post-dose Period 1
Description: Vz/F is the distribution of study drug between the plasma and the rest of the body after the dose. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail in healthy participants, participants with renal impairment, and 24 hours prior to hemodialysis in participants with end-stage renal disease requiring hemodialysis. Vz/F was to be calculated for the parent plasma analytes only, midazolam, dabigatran, pitavastatin, atorvastatin, and rosuvastatin.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose
Population: All participants who were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of Vz/F for the following reasons: non-compliance with the protocol or high pre-dose concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | End-Stage Renal Disease | Severe Impairment | Moderate Impairment | Mild Impairment | Healthy Control
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6
liters
  Midazolam | 579 (45.0) | 433 (16.9) | 409 (38.0) | 555 (58.0) | 422 (37.5)
  Dabigatran: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
  Dabigatran | 3140 (38.4) | 1230 (36.4) | 1060 (54.1) | 2120 (57.9) | 1730 (46.4)
  Pitavastatin | 252 (19.5) | 454 (51.9) | 317 (15.4) | 405 (46.8) | 495 (46.6)
  Atorvastatin: number analyzed (Participants) | 6 | 7 | 6 | 4 | 6
  Atorvastatin | 3520 (40.3) | 5310 (47.7) | 5240 (57.5) | 7300 (32.5) | 7380 (58.6)
  Rosuvastatin: number analyzed (Participants) | 5 | 6 | 5 | 4 | 3
  Rosuvastatin | 4870 (63.2) | 3720 (51.3) | 3120 (35.9) | 4270 (117.9) | 4010 (34.4)

11. Secondary Outcome: Effect of Rifampin on AUC0-24 Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the AUC0-24 of midazolam, dabigatran, pitavastatin, pitavastatin lactone, atorvastatin, ortho-hydroxyatorvastatin, and rosuvatatin. AUC0-24 is the area under the plasma concentration-time curve from time 0 to 24 hours post-dose. This is a measure of the average amount of study drug in the blood plasma over a period of 24 hours after the dose. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: Microdose cocktail: 0 hour (pre-dose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose; rifampin: 0 hour (pre-dose) and 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 24 hours post-dose
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of AUC0-24 for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg*hr/mL
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
pg*hr/mL
  Midazolam |  | 238 [171 to 330] | 346 [224 to 490] | 186 [131 to 263] | 234 [165 to 332]
  Dabigatran |  | 6540 [4730 to 9030] | 5480 [3900 to 7700] | 2660 [1890 to 3740] | 3030 [2160 to 4260]
  Pitavastatin |  | 2760 [1780 to 4270] | 3360 [2120 to 5330] | 2460 [1550 to 3900] | 1860 [1170 to 2950]
  Pitavastatin lactone (metabolite) |  | 1070 [820 to 1400] | 1780 [1340 to 2350] | 1490 [1120 to 1970] | 1000 [755 to 1320]
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 2230 [1510 to 3290] | 2420 [1610 to 3630] | 1700 [1030 to 2790] | 1760 [1180 to 2650]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) |  | 1580 [1060 to 2350] | 1800 [1190 to 2730] | 1720 [1030 to 2870] | 1620 [1070 to 2460]
  Rosuvastatin: number analyzed (Participants) | 0 | 6 | 6 | 5 | 6
  Rosuvastatin |  | 1100 [779 to 1550] | 1670 [1170 to 2400] | 1010 [682 to 1500] | 842 [588 to 1210]

12. Secondary Outcome: Effect of Rifampin on AUC0-last Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the AUC0-last of midazolam, dabigatran, pitavastatin, pitavastatin lactone, atorvastatin, ortho-hydroxyatorvastatin, and rosuvatatin. AUC0-last is the area under the plasma concentration-time curve from time zero to time of last measurable concentration. It is a measure of the amount of study drug in the blood plasma from pre-dose until the last measurable concentration of study drug could be determined. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: as for outcome 2
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of AUC0-last for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg*hr/mL
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
pg*hr/mL
  Midazolam |  | 236 [168 to 331] | 353 [246 to 505] | 182 [127 to 261] | 231 [161 to 331]
  Dabigatran |  | 10400 [7310 to 14800] | 6830 [4710 to 9920] | 2830 [1950 to 4110] | 3140 [2160 to 4550]
  Pitavastatin |  | 2850 [1830 to 4430] | 3480 [2180 to 5540] | 2510 [1580 to 4000] | 1890 [1190 to 3010]
  Pitavastatin lactone (metabolite) |  | 1470 [1100 to 1980] | 2380 [1750 to 3250] | 1850 [1350 to 2520] | 1270 [935 to 1740]
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 2220 [1490 to 3290] | 2420 [1600 to 3650] | 1690 [1020 to 2800] | 1760 [1160 to 2650]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) |  | 1610 [1080 to 2400] | 1850 [1220 to 2820] | 1750 [1050 to 2920] | 1630 [1070 to 2470]
  Rosuvastatin: number analyzed (Participants) | 0 | 6 | 6 | 5 | 6
  Rosuvastatin |  | 1150 [806 to 1630] | 1740 [1200 to 2500] | 1040 [698 to 1560] | 854 [592 to 1230]

13. Secondary Outcome: Effect of Rifampin on Cmax Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the Cmax of midazolam, dabigatran, pitavastatin, pitavastatin lactone, atorvastatin, ortho-hydroxyatorvastatin, and rosuvatatin. Cmax is the peak plasma concentration of study drug after administration. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: Microdose cocktail: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 32, 48, and 72 hours post-dose; rifampin: 0.5, 1, 1.5, 2, 3, 4, 6, 12, and 24 hours post-dose
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of Cmax for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
pg/mL
  Midazolam |  | 75.4 [57.1 to 99.7] | 92.5 [69.0 to 124] | 73.0 [54.5 to 97.9] | 81.4 [60.7 to 109]
  Dabigatran |  | 422 [305 to 584] | 443 [314 to 624] | 243 [173 to 342] | 351 [249 to 494]
  Pitavastatin |  | 981 [591 to 1630] | 860 [509 to 1450] | 819 [485 to 1380] | 599 [354 to 1010]
  Pitavastatin lactone (metabolite) |  | 88.4 [72.8 to 107] | 119 [97.3 to 145] | 131 [108 to 161] | 102 [83.7 to 125]
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 531 [354 to 796] | 508 [337 to 766] | 505 [305 to 835] | 405 [269 to 611]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) |  | 150 [97.1 to 231] | 174 [111 to 272] | 215 [124 to 372] | 198 [126 to 310]
  Rosuvastatin: number analyzed (Participants) | 0 | 6 | 6 | 5 | 6
  Rosuvastatin |  | 208 [133 to 327] | 396 [248 to 633] | 254 [152 to 425] | 236 [148 to 376]

14. Secondary Outcome: Effect of Rifampin on C24 Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the C24 of midazolam, dabigatran, pitavastatin, pitavastatin lactone, atorvastatin, ortho-hydroxyatorvastatin, and rosuvatatin. C24 is a measure of the plasma study drug concentration 24 hours post-dose. C24 is reported as median (minimum and maximum) in severe renal impairment arm due to zero values. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: 24 hours post-dose
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of C24 for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
pg/mL
  Midazolam |  | 0.394 [0.00 to 4.15] | 1.42 [0.701 to 2.89] | 0.00 [0.00 to 0.921] | 0.601 [0.00 to 1.33]
  Dabigatran |  | 174 [115 to 263] | 100 [65.1 to 154] | 31.1 [20.2 to 47.9] | 27.5 [17.9 to 42.4]
  Pitavastatin |  | 7.01 [3.81 to 12.9] | 10.5 [5.54 to 19.8] | 4.70 [2.49 to 8.87] | 4.72 [2.50 to 8.91]
  Pitavastatin lactone (metabolite) |  | 21.3 [15.0 to 30.3] | 34.0 [23.5 to 49.3] | 20.7 [14.3 to 30.0] | 17.1 [11.8 to 24.8]
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 2.98 [0.00 to 16.1] | 2.98 [1.65 to 5.40] | 1.76 [0.00 to 2.32] | 1.35 [0.00 to 3.20]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) |  | 7.23 [3.70 to 14.1] | 9.96 [5.02 to 19.8] | 6.28 [2.71 to 14.5] | 5.57 [2.81 to 11.1]
  Rosuvastatin: number analyzed (Participants) | 0 | 6 | 6 | 5 | 6
  Rosuvastatin |  | 4.47 [2.34 to 8.53] | 6.97 [3.53 to 13.8] | 4.18 [1.22 to 9.99] | 2.42 [0.00 to 6.92]

15. Secondary Outcome: Effect of Rifampin on Tmax Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the Tmax of midazolam, dabigatran, pitavastatin, pitavastatin lactone, atorvastatin, ortho-hydroxyatorvastatin, and rosuvatatin. Tmax is the amount of time to reach maximum (peak) plasma drug concentration following drug administration. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: as for outcome 13
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of Tmax for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Median (Full Range); unit: hours
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
hours
  Midazolam |  | 0.50 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 0.50 [0.50 to 1.00] | 1.00 [0.50 to 1.00]
  Dabigatran |  | 3.50 [2.00 to 4.05] | 3.00 [2.00 to 4.00] | 2.50 [2.00 to 4.00] | 2.50 [1.50 to 3.00]
  Pitavastatin |  | 1.00 [0.50 to 1.00] | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 3.00] | 1.00 [1.00 to 2.00]
  Pitavastatin lactone (metabolite) |  | 3.00 [1.50 to 4.00] | 4.00 [2.00 to 12.00] | 3.00 [1.50 to 4.00] | 2.00 [1.50 to 4.05]
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 0.50 [0.50 to 1.00] | 1.50 [0.50 to 2.00] | 1.00 [1.00 to 1.50] | 1.50 [1.00 to 2.00]
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) |  | 1.75 [1.00 to 4.05] | 2.50 [1.50 to 4.00] | 1.75 [1.00 to 4.00] | 3.00 [1.00 to 4.05]
  Rosuvastatin: number analyzed (Participants) | 0 | 6 | 6 | 5 | 6
  Rosuvastatin |  | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 2.00 [1.00 to 6.00]

16. Secondary Outcome: Effect of Rifampin on t1/2 Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the t1/2 of midazolam, dabigatran, pitavastatin, pitavastatin lactone, atorvastatin, ortho-hydroxyatorvastatin, and rosuvatatin. T1/2 is the elimination half-life of study drug. T1/2 is the time it takes for half of the study drug in the blood plasma to dissipate. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: as for outcome 13
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of t1/2 for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
hours
  Midazolam |  | 4.14 (19.5) | 5.49 (26.2) | 4.12 (26.7) | 4.97 (22.0)
  Dabigatran |  | 19.4 (21.3) | 11.3 (33.1) | 7.57 (19.0) | 6.48 (13.7)
  Pitavastatin |  | 6.99 (62.8) | 11.5 (71.6) | 8.40 (75.8) | 6.50 (30.3)
  Pitavastatin lactone (metabolite) |  | 17.2 (41.0) | 17.7 (25.2) | 21.0 (22.5) | 16.5 (33.9)
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 3.14 (18.9) | 2.99 (21.1) | 3.22 (8.6) | 2.76 (8.4)
  Ortho-hydroxyatorvastatin (metabolite): number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Ortho-hydroxyatorvastatin (metabolite) |  | 4.56 (43.7) | 4.25 (39.7) | 3.83 (19.7) | 3.49 (11.7)
  Rosuvastatin: number analyzed (Participants) | 0 | 5 | 4 | 5 | 5
  Rosuvastatin |  | 4.89 (49.9) | 7.48 (19.8) | 9.64 (83.8) | 6.76 (94.3)

17. Secondary Outcome: Effect of Rifampin on CL/F Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the CL/F of midazolam, dabigatran, pitavastatin, atorvastatin, and rosuvatatin. CL/F is the rate at which study drug was removed from the body. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: as for outcome 13
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of CL/F for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
liters/hour
  Midazolam |  | 40.5 (57.7) | 27.8 (52.0) | 53.0 (34.8) | 41.8 (28.4)
  Dabigatran |  | 26.3 (41.6) | 38.9 (58.7) | 92.8 (41.5) | 85.6 (40.0)
  Pitavastatin |  | 3.57 (50.0) | 2.86 (60.4) | 3.95 (51.8) | 5.24 (75.8)
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 44.2 (57.6) | 41.1 (30.3) | 58.6 (49.4) | 56.4 (62.2)
  Rosuvastatin: number analyzed (Participants) | 0 | 5 | 4 | 5 | 5
  Rosuvastatin |  | 38.6 (37.7) | 28.9 (41.1) | 47.1 (51.1) | 57.9 (63.3)

18. Secondary Outcome: Effect of Rifampin on Vz/F Post-dose Period 2
Description: To evaluate the effect of a single oral dose of rifampin on the Vz/F of midazolam, dabigatran, pitavastatin, pitavastatin lactone, atorvastatin, ortho-hydroxyatorvastatin, and rosuvatatin. Vz/F is the distribution of study drug between the plasma and the rest of the body after the dose. Plasma pharmacokinetic data presented in the table below are following the administration of a single oral dose of a microdose cocktail and rifampin in healthy participants and participants with renal impairment. As pre-specified in the protocol, this outcome measure does not include end-stage renal disease participants as they did not receive rifampin during Period 2.
Time Frame: as for outcome 13
Population: All participants who received rifampin, were compliant with the study procedure and had available data. Per protocol, participants were excluded from this analysis of Vz/F for the following reasons: non-compliance with the protocol or high pre-dose concentrations. Per protocol, end-stage renal disease participants did not receive rifampin.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | End Stage Renal Disease (Period 2) | Severe Impairment (Period 2) | Moderate Impairment (Period 2) | Mild Impairment (Period 2) | Healthy Control (Period 2)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6
liters
  Midazolam |  | 242 (44.6) | 220 (56.5) | 315 (30.8) | 300 (36.3)
  Dabigatran |  | 733 (29.2) | 632 (36.3) | 1010 (45.2) | 800 (41.1)
  Pitavastatin |  | 36.0 (38.7) | 47.3 (85.8) | 47.8 (82.5) | 49.2 (72.1)
  Atorvastatin: number analyzed (Participants) | 0 | 6 | 6 | 4 | 6
  Atorvastatin |  | 200 (55.4) | 177 (38.2) | 272 (58.4) | 225 (68.7)
  Rosuvastatin: number analyzed (Participants) | 0 | 5 | 4 | 5 | 5
  Rosuvastatin |  | 272 (39.7) | 313 (58.2) | 654 (40.8) | 565 (76.1)

ADVERSE EVENTS:
Time Frame: Up tp approximately 30 days (including 14 days following the last dose)
Description: All participants who received any dose are included. Adverse events were summarized by renal function group assignment and dose received (microdose cocktail alone or microdose cocktail + rifampin).
Groups:
- End Stage Renal Disease: Microdose Cocktail Alone: Participants requiring hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution).
  Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). A washout period of at least 14 days will separate dosings.
- Severe Impairment: Microdose Cocktail Alone: Participants with <30 mL/min/1.73m^2 eGFR not on hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution).
- Severe Impairment: Microdose Cocktail + Rifampin: Participants with <30 mL/min/1.73m^2 eGFR not on hemodialysis. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
- Moderate Impairment: Microdose Cocktail Alone: Participants with 30 to <60 mL/min/1.73m^2 eGFR not on hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution).
- Moderate Impairment: Microdose Cocktail + Rifampin: Moderate ImpairmentEdit Participants with 30 to <60 mL/min/1.73m^2 eGFR not on hemodialysis. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
- Mild Impairment: Microdose Cocktail Alone: Participants with 60 to <90 mL/min/1.73m^2 eGFR not on hemodialysis. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution).
- Mild Impairment: Microdose Cocktail + Rifampin: Participants with 60 to <90 mL/min/1.73m^2 eGFR not on hemodialysis. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
- Healthy Control: Microdose Cocktail Alone: Participants with ≥90 mL/min creatinine clearance. Period 1/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution). Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
- Healthy Control: Microdose Cocktail + Rifampin: Participants with ≥90 mL/min creatinine clearance. Period 2/Day 1: participants receive a single oral dose of the microdose cocktail (midazolam oral solution, dabigatran etexilate and pitavastatin oral solution, atorvastatin and rosuvastatin oral solution) and rifampin. A washout period of at least 14 days will separate dosings.
Arm/Group | End Stage Renal Disease: Microdose Cocktail Alone | Severe Impairment: Microdose Cocktail Alone | Severe Impairment: Microdose Cocktail + Rifampin | Moderate Impairment: Microdose Cocktail Alone | Moderate Impairment: Microdose Cocktail + Rifampin | Mild Impairment: Microdose Cocktail Alone | Mild Impairment: Microdose Cocktail + Rifampin | Healthy Control: Microdose Cocktail Alone | Healthy Control: Microdose Cocktail + Rifampin
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 2/7 | 1/6 | 2/6 | 1/6 | 3/7 | 2/6 | 0/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | End Stage Renal Disease: Microdose Cocktail Alone (N=6) | Severe Impairment: Microdose Cocktail Alone (N=7) | Severe Impairment: Microdose Cocktail + Rifampin (N=6) | Moderate Impairment: Microdose Cocktail Alone (N=6) | Moderate Impairment: Microdose Cocktail + Rifampin (N=6) | Mild Impairment: Microdose Cocktail Alone (N=7) | Mild Impairment: Microdose Cocktail + Rifampin (N=6) | Healthy Control: Microdose Cocktail Alone (N=6) | Healthy Control: Microdose Cocktail + Rifampin (N=6)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | End Stage Renal Disease: Microdose Cocktail Alone (N=6) | Severe Impairment: Microdose Cocktail Alone (N=7) | Severe Impairment: Microdose Cocktail + Rifampin (N=6) | Moderate Impairment: Microdose Cocktail Alone (N=6) | Moderate Impairment: Microdose Cocktail + Rifampin (N=6) | Mild Impairment: Microdose Cocktail Alone (N=7) | Mild Impairment: Microdose Cocktail + Rifampin (N=6) | Healthy Control: Microdose Cocktail Alone (N=6) | Healthy Control: Microdose Cocktail + Rifampin (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will provide separate guidance on the criteria for publication of clinical trial data when contacted for permission to publish.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03311841/Prot_SAP_000.pdf